CLINICAL TRIAL: NCT06539286
Title: Dentin Hypersensitivity - Varnish or Laser? A Randomized Clinical Study Comparing Three Wavelengths (2940 nm, 1064 nm and 970 nm) and the Desensitizer Gluma
Brief Title: Dentin Hypersensitivity - Varnish or Laser?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DH
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will not know which laser will be used in the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): Desensitizing Agent Gluma
  Interventions: Device: Laser Irradiation
- 1. Laser Group (Active Comparator): Er:YAG laser
  Interventions: Device: Laser Irradiation
- 2. Laser Group (Active Comparator): Nd:YAG laser
  Interventions: Device: Laser Irradiation
- 3. Laser Group (Active Comparator): 970 nm diode laser
  Interventions: Device: Laser Irradiation

INTERVENTIONS:
Device: Laser Irradiation — three different laser wavelengths will be used
  Other Names: Desensitizing Agent Gluma

SUMMARY:
Dentin hypersensitivity is a common condition described as a short and sharp pain caused by thermal, evaporative, tactile, osmotic, or chemical stimuli to exposed dentin that cannot be related to another defect or dental pathology. The variety of treatment options and products on the market might seem overwhelming. This study aims to show that laser treatments are efficient in reducing pain scores compared to a desensitizing agent (Gluma). 80 patients with at least two hypersensitive teeth will be enrolled in this study. Patients will be divided randomly into four groups (control group (Gluma), laser group 1 (2.94 µm wavelength), laser group 2 (1064 nm wavelength), laser group 3 (970 nm wavelength)). Visual Analog Scale will be measured before treatment, right after treatment, one week after treatment, one month after treatment, three months after treatment. Mixed Anova's and descriptive analysis will be used for statistical evaluation.

DETAILED DESCRIPTION:
A total of 80 patients meeting the inclusion criteria will be included in this randomized clinical study. Participants will be randomly divided into four groups. Pain scores will be measured before treatment, right after treatment, 1 month after treatment and 3 months after treatment using the Visual Analog Scala (VAS). Patients will not know which treatment will be performed before nor will the patients from the laser groups know the wavelengths. Pain scores at check-up meetings will be collected by another doctor other than the one who will perform all laser treatments.

ELIGIBILITY:
Inclusion Criteria:

* all genders
* 18-70 years
* good general health
* at least two hypersensitive teeth in either jaw
* initial VAS-score >3

Exclusion Criteria:

* Active carious lesions, insufficient restorations, enamel cracks, reversible pulpitis
* Active periodontal disease, periodontal surgery (in the last 6 months)
* Bleaching procedure in the last 3 months
* Analgetic use in the last 72 hours
* Pregnant/lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2024-10-14 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale changes | three months
  Patients will rate pain score with VAS. Pain scores will be evaluated before treatment, right after treatment, one week later, one month later and three months later